CLINICAL TRIAL: NCT07015775
Title: Evaluation of the Analgesic Efficacy of an Ultrasound-guided Transperineal Pudendal Block in Outpatient Hemorrhoidal Surgery
Acronym: BACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-A00534-45
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hemorrhoids
Keywords: hemorroidal surgery
MeSH Terms: conditions — Hemorrhoids | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, randomized, double-blind study conducted on two parallel groups of patients undergoing hemorrhoidal surgery (pudendal block guided by neurostimulation versus pudendal block guided by ultrasound).
Who Masked: Participant, Investigator
Masking Description: To maintain double blinding, postoperative data will be collected by a physician other than the anesthesiologist performing the block, and by nursing staff under their supervision. None of these personnel will be informed of the patient's group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block guided by neurostimulation (Active Comparator): Neurostimulation involves using an electrical impulse to trigger a nerve signal and a specific motor response. A short-bevel, insulated 80 mm needle connected to a neurostimulator is used. The puncture point lies midway between the ischial tuberosity and the anus. Stimulation starts at 2.5 mA, 1 Hz, and the needle is advanced 4-5 cm until anal sphincter contraction occurs ("anal wink"). The needle is adjusted to maintain the response while reducing intensity to 0.5 mA. If lost, intensity is increased; if too intense at 0.3 mA, the needle is repositioned. After confirming no vascular puncture, 1 mL of Ropivacaine 3.5 mg/mL is injected to stop contraction, followed by slow injection of 15 mL total. The procedure is repeated on the other side. If no motor response occurs, a blind injection is performed after negative aspiration at 5 cm depth using the same landmarks.
  Interventions: Procedure: Neurostimulation
- Pudendal block guided by ultrasound (Experimental): A 6 MHz convex probe is placed in the frontal plane along the line between the ischial tuberosity and the anal margin to visualize the bony prominence. The pudendal artery and nearby nerves are identified using color Doppler. A 22-gauge, 80 mm echogenic needle is inserted out-of-plane in front of the probe, targeting the lateral ischioanal fossa just medial to the pudendal artery, if visible. The probe is adjusted to center the artery. Block confirmation is based on ultrasound visualization of local anesthetic spreading into the fatty tissue medial to the pudendal artery. The procedure is repeated on the other side. If the artery is not visible, the injection is performed after negative aspiration on the medial aspect of the ischial tuberosity, along the line to the anus, at a depth of 4-5 cm.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Neurostimulation — Procedure guided by neurostimulation
  Arms: Pudendal block guided by neurostimulation
Procedure: Ultrasound — Procedure guided by ultrasound
  Arms: Pudendal block guided by ultrasound

SUMMARY:
In a population of patients undergoing hemorrhoidal surgery under general anesthesia and divided into two equal groups based on the method used for intraoperative pudendal nerve block and its branches in the ischioanal fossa:

Group 1: Pudendal block guided by neurostimulation Group 2: Pudendal block guided by ultrasound

The primary objective of this study is to compare the maximum immediate postoperative pain score between the two groups (pain reported by the patients in the recovery room on a simple numeric scale before morphine titration).

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind study conducted on two parallel groups of patients undergoing hemorrhoidal surgery (pudendal block guided by neurostimulation versus pudendal block guided by ultrasound).

Study Duration The total study duration per patient is 7 days. The recruitment period is set at 12 months.

Justification of the Experimental Protocol The aim of this study is to compare two methods of performing a pudendal block. Patient allocation to either strategy will be determined by randomization. Bilateral pudendal nerve block and its branches in the ischioanal fossa will be performed after induction of general anesthesia.

To maintain double blinding, postoperative data will be collected by a physician other than the anesthesiologist performing the block, and by nursing staff under their supervision. None of these personnel will be informed of the patient's group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient
* Patient who has signed informed consent to participate in the study
* Patient scheduled for outpatient hemorrhoidal surgery under general anesthesia

Exclusion Criteria:

* History of hemorrhoidal surgery
* Allergy or contraindication to any of the medications used in the study
* Patient undergoing surgery under spinal anesthesia
* History of chronic pain requiring opioid use, unrelated to hemorrhoids
* Mental impairment or any other condition that could hinder understanding or strict adherence to the protocol
* Patient not affiliated with the French national health insurance system
* Patient under legal protection (e.g., guardianship, trusteeship, or court protection)
* Pregnant woman or woman at risk of being pregnant (i.e., of childbearing age without effective contraception and without an HCG test)
* Patient already enrolled in another therapeutic clinical trial or within the exclusion period of another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain assessment in the Post-Anesthesia Care Unit (PACU) | Hour 2
  The primary endpoint of the study is the maximum pain score in the Post-Anesthesia Care Unit (PACU) before morphine titration.
  Postoperative pain in the recovery room will be recorded by the nursing staff using a simple numeric scale from 0 to 10 after questioning the patient, following standard departmental procedures. The maximum pain score before morphine titration constitutes the primary evaluation criterion.

SECONDARY OUTCOMES:
Quantitative Opioid Consumption | Hour 2
  Mean amount of morphine administered in each group
Qualitative Opioid Consumption | Hour 2
  Percentage of patients in each group with zero morphine use
Postoperative recovery assessment | Day 1
  QOR-15 accurately assesses postoperative recovery across five key domains: pain, physical comfort, physical independence, psychological support, and emotional state. Each item is rated from 0 (poor) to 10 (excellent), with a total score ranging from 0 (no recovery) to 150 (full recovery).
Postoperative recovery assessment | Day 3
  QOR-15 accurately assesses postoperative recovery across five key domains: pain, physical comfort, physical independence, psychological support, and emotional state. Each item is rated from 0 (poor) to 10 (excellent), with a total score ranging from 0 (no recovery) to 150 (full recovery).
Postoperative recovery assessment | Day 7
  QOR-15 accurately assesses postoperative recovery across five key domains: pain, physical comfort, physical independence, psychological support, and emotional state. Each item is rated from 0 (poor) to 10 (excellent), with a total score ranging from 0 (no recovery) to 150 (full recovery).
Postoperative Pain assessment at rest | Day 1
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Postoperative Pain assessment at rest | Day 3
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Postoperative Pain assessment at rest | Day 7
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Postoperative Pain assessment during walking | Day 1
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Postoperative Pain assessment during walking | Day 3
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Postoperative Pain assessment during walking | Day 7
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Postoperative Pain assessment during First defecation | Day 7
  Postoperative pain will be measured by nursing staff during the patient's ambulatory stay, and the maximum score will be recorded in the Case Report Form (CRF). Pain will be self-reported by the patient using a simple numeric scale from 0 to 10.
Non-Opioid Postoperative Medication Use | Day 1
  Use of non-opioid analgesics and antiemetics during hospitalization. Use of analgesics as reported by the patients.
Pudendal block procedure duration | Hour 2
  Duration of pudendal block procedure
Sensory block duration | Day 7
  Duration of sensory block
Length of stay in the PACU | Day 1
  Length of stay in the PACU
Total hospital stay duration | Day 1
  Total hospital stay duration
Time to first defecation | Day 7
  Time to first defecation
Tolerance | Day 7
  Procedure tolerance will be assessed by recording all adverse events (serious or non-serious) with a potential causal link to analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas GIRAL, MD, Principal Investigator — Hôpital privé Claude Galien
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France

REFERENCES:
- [Derived] Giral T, Maupain O, Elmaleh Y, Huynh D, Ciceron F, Yao K, Devidas P, El Metni A, Kutter J. Ultrasound-guided versus neurostimulation-guided bilateral transperineal pudendal nerve block for analgesia in outpatient haemorrhoid surgery: protocol for a multicentre, randomised, double-blind, non-inferiority trial. BJA Open. 2025 Dec 9;16:100512. doi: 10.1016/j.bjao.2025.100512. eCollection 2025 Dec. PMID 41476689